CLINICAL TRIAL: NCT07300462
Title: A Randomized, Double-blind, Placebo-Controlled Clinical Study to Evaluate the Protective Efficacy of Oral Recombinant Subunit B/Bacterial Cholera Vaccine (Enteric-coated Capsules) Against Infectious Diarrhea Caused by Non-Vibrio Cholerae in Healthy People Aged 2 to 14 Years
Brief Title: A Post-marketing Observational Study of Oral Cholera Vaccine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai United Cell Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OCV-YJFA-2024-001
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diarrhea
Keywords: IV
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules) (Experimental)
  Interventions: Biological: Recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules)
- Recombinant B subunit/bacterial cholera vaccine (enteric-coated capsule) placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules) — The participants in the experimental group will be given three oral doses of recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules) on D0, D7, and D28 .
  Arms: Recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules)
Biological: Placebo — The participants in the Control group will be given three oral doses of recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules) Placebo on D0, D7, and D28 .
  Arms: Recombinant B subunit/bacterial cholera vaccine (enteric-coated capsule) placebo

SUMMARY:
Chinese survey data indicate that the incidence rate of diarrhea in the general population ranges from 0.17 to 0.70 episodes per person-year, whereas among children under five years of age, the rate is significantly higher, ranging from 2.50 to 3.38 episodes per person-year. Over recent decades, rapid economic development has contributed substantially to the reduction of mortality associated with infectious diseases. However, emerging challenges-such as increasing antimicrobial resistance and heightened population mobility-have complicated efforts in infectious disease prevention and control. In a phase III clinical trial of the recombinant B subunit/bacterial whole-cell cholera vaccine (enteric-coated capsule), a statistically significant difference was observed in the overall incidence of diarrhea between the vaccinated group (12.9%) and the control group (26.7%) (P < 0.01). Findings from similar vaccine studies conducted in Sweden have demonstrated cross-protection against diarrhea caused by enterotoxigenic Escherichia coli (ETEC) and other intestinal pathogens. Specifically, the vaccine conferred a 50% protection rate against Salmonella enterica infections, 82% against mixed infections involving ETEC and Salmonella, and 71% against mixed infections involving ETEC and other pathogens. Evidence from relevant studies suggests that the recombinant B subunit/bacterial whole-cell cholera vaccine may offer protective benefits against non-cholera infectious diarrhea. Nevertheless, there remains a paucity of real-world effectiveness data, particularly in pediatric populations who bear a disproportionately high burden of diarrheal disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 years old, ≤ 14 years old, male or female.
2. Not vaccinated against cholera.
3. Obtain the consent of the study subject or guardian and sign the informed consent form.
4. The subjects and their guardians were able to comply with the requirements of the clinical study protocol.
5. Axillary temperature < 37.0 °C was measured on the day of inoculation.

Exclusion Criteria:

* Exclusion Criteria for First Inoculation：

  1. Patients with febrile illness (axillary temperature ≥ 37.0 °C on the day of vaccination), other acute diseases, and diarrhea within 7 days before vaccination.
  2. Use of antibiotics within 7 days prior to vaccination.
  3. Patients with gastric ulcer, abnormal gastric acid secretion and other gastric diseases or discomfort.
  4. History of allergy to vaccinations and oral medications.
  5. Patients with congenital malformations, developmental disorders, or severe chronic diseases.
  6. Suspected progressive neurological disorder, epilepsy, or long-term use of antibiotics.
  7. Received blood products within 3 months prior to vaccination.
  8. Received other investigational drugs within 30 days prior to vaccination.
  9. Received any Rotavirus vaccine within 12 months prior to vaccination.
  10. Live attenuated vaccine within 14 days or subunit or inactivated vaccine within 7 days prior to vaccination.
  11. Asthma requiring urgent treatment, hospitalization, intubation, oral or intravenous corticosteroids for unstable past two years.
  12. Patients with severe hypertension, heart, liver, kidney disease, and severe infectious diseases (acquired immunodeficiency syndrome and active tuberculosis).
  13. Has a malignancy, is active or has been treated without definitive cure, or has the potential to relapse during the study.
  14. Epilepsy, excluding epilepsy that has been discontinued within the past 3 years and has not recurred.
  15. Patients with coagulation disorders.
  16. Those who have had or are currently suffering from mental illness that have not been well controlled within the past two years due to psychological conditions that do not comply with protocol requirements, and who need to take drugs for psychosis.
  17. In the judgment of the investigator, it is contrary to the protocol due to various medical, psychological, social or other conditions, or affects the subject to sign the informed consent.
* Exclusion Criteria for Second and Third Oral Vaccines：

  1. Those who have an allergic reaction at the time of the first or second vaccination.
  2. Occurring in any of the first dose exclusion criteria after inclusion.
  3. Serious adverse event causally related to first or second dose of study vaccine.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 6000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of infectious diarrhea in the vaccinated group and placebo group | The incidence of diarrhea in the experimental group and the control group within 180 days starting from 7 days after full immunization (the baseline day for diarrhea)
  Protective effect of recombinant subunit B/bacterial cholera vaccine (enteric-coated capsules) against infectious diarrhea due to enteropathogens (except Vibrio cholerae) (Day 7 after full immunization to the end of the study).

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anhui Provincial Center for Disease Control and Prevention, Hefei, Anhui
  - National Institute for Communicable Disease Control and Prevention, China, Beijing, Beijing Municipality
  - Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei
  - Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu
  - Shandong Provincial Center for Disease Control and Prevention, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No